CLINICAL TRIAL: NCT04525261
Title: Natural History of Patients With Inherited Retinal Diseases Due to Mutations in RPE65 Gene
Acronym: RPE65-NHS
Status: Completed | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Retina Italia Onlus (Unknown)
Responsible Party: Principal Investigator, Francesca Simonelli, Prof, University of Campania Luigi Vanvitelli
Other Study IDs: RPE65-NHS
Record Dates: First submitted 2020-07-31; First posted 2020-08-25 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Leber Congenital Amaurosis 2; Retinitis Pigmentosa 20
Keywords: RPE65-related inherited retinal dystrophies; natural history study
MeSH Terms: conditions — Amaurosis congenita of Leber, type 2; Retinitis Pigmentosa 20

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale:

In preparation for treatment with gene therapy, this study is being conducted in order to investigate the natural history of Inherited Retinal Dystrophies (IRDs) due to mutations in RPE65 gene. Such a study will help identify suitable patients for therapeutic intervention.

Methodology:

This is a multicenter retrospective, descriptive chart review study designed to assess retinal structure and function in subjects with IRDs due to mutation in RPE65 gene by visual acuity, visual field measurements, Optical Coherence Tomography (OCT), and a number of other vision-related assessments.

ELIGIBILITY:
Inclusion Criteria:

* Must be willing to adhere to protocol as evidenced by written informed consent or parental permission and subject assent.
* Subjects diagnosed with Retinitis Pigmentosa or Leber Congenital Amaurosis.
* Molecular diagnosis showing mutations (homozygotes or compound heterozygotes) in RPE65 gene.
* Age three years old or older.
* Minimum of two office / clinic visits encounters with ophthalmic assessment that span a follow-up period of at least 1 year with the last visit occurring within the last six months (before signature of informed consent and of study start).

Exclusion Criteria:

* Unable or unwilling to meet requirements of the study.
* Participation in a clinical study with an investigational drug during the retrospective study time period (i.e., from 01/01/1990 to study start date).

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: It is expected that approximately 200 patients may be recruited into the study during the recruitment period.
  Each subject must participate in the informed consent process and provide written informed consent/assent before any data could be collected.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
best correct visual acuity | at least one year
  average annual progression rate of best correct visual acuity over the retrospective follow-up period
visual field | at least one year
  average annual progression rate of visual field over the retrospective follow-up period
optical coherence tomography | at least one year
  average annual progression rate of central retinal thickness over the retrospective follow-up period

SECONDARY OUTCOMES:
microperimetry | at least one year
  average annual progression rate of macular sensitivity assessed by microperimetry over the retrospective follow-up period
fundus autofluorescence | at least one year
  change in fundus autofluorescence over the retrospective follow-up period
Full-field Electroretinogram | at least one year
  average annual progression rate of full-field electroretinogram responses over the retrospective follow-up period
Multifocal Electroretinogram | at least one year
  average annual progression rate of multifocal electroretinogram responses over the retrospective follow-up period

CONTACTS AND LOCATIONS:
Locations (9):
- Italy (9):
  - Ospedale di Camposampiero, ULSS6 Euganea, Camposampiero, Camposampiero
  - UOC Oculistica - AOU Careggi, Florence
  - UOC Oculistica - Ospedale Sacco, Milan
  - UOC Oculistica - Ospedale San Paolo, Milan
  - UOC Oculistica - AOU Università degli Studi della Campania Luigi Vanvitelli, Naples
  - Centro di Neuroftalmologia dell'età evolutiva - IRCCS Fondazione Istituto Neurologico Nazionale C. Mondino, Pavia
  - UOC Oculistica - Fondazione IRCCS Policlinico San Matteo, Pavia
  - UOC Oculistica - Ospedale Bambin Gesù di Roma, Rome
  - UOC Oculistica - Policlinico Gemelli di Roma, Rome

IPD SHARING:
Plan to Share IPD: No